CLINICAL TRIAL: NCT06682351
Title: Heterogeneity of Diabetes: Integrated Muli-Omics to Identify Physiologic Subphenotypes and Evaluate Targeted Prevention
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Tracey McLaughlin, Professor of Medicine (Endocrinology), Stanford University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 76481
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Prediabetes / Type 2 Diabetes
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2 | interventions — Metformin; glucagon-like peptide 1 (7-36)amide; Glucagon-Like Peptide 1; Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Mediterranean Diet/GLP1a/Metformin (Experimental): 1. 16 weeks of following a Mediterranean diet: a mostly plant-based diet that includes vegetables, whole grains, whole fruits, legumes, nuts and seeds, with fish being the primary animal protein, and olive oil the primary fat.
  2. 3 months washout
  3. 16 weeks using GLP1 agonist: Dosing will be titrated per clinical guidelines and as per FDA approved clinical protocols.
  4. 3 months washout
  5. 16 weeks of using metformin: Dosing will initiate at 500mg TID and increased to 1000mg BID after one week.
  Interventions: Drug: Metformin; Drug: GLP-1A; Dietary Supplement: MED
- Metformin/Mediterranean Diet/GLP1a (Experimental): 1. 16 weeks of using metformin: Dosing will initiate at 500mg TID and increased to 1000mg BID after one week.
  2. 3 months washout
  3. 16 weeks of following a Mediterranean diet: a mostly plant-based diet that includes vegetables, whole grains, whole fruits, legumes, nuts and seeds, with fish being the primary animal protein, and olive oil the primary fat.
  4. 3 months washout
  5. 16 weeks using GLP1 agonist: Dosing will be titrated per clinical guidelines and as per FDA approved clinical protocols.
  Interventions: Drug: Metformin; Drug: GLP-1A; Dietary Supplement: MED
- GLP1a/Metformin/Mediterranean Diet (Experimental): 1. 16 weeks using GLP1 agonist: Dosing will be titrated per clinical guidelines and as per FDA approved clinical protocols.
  2. 3 months washout
  3. 16 weeks of using metformin: Dosing will initiate at 500mg TID and increased to 1000mg BID after one week.
  4. 3 months washout
  5. 16 weeks of following a Mediterranean diet: a mostly plant-based diet that includes vegetables, whole grains, whole fruits, legumes, nuts and seeds, with fish being the primary animal protein, and olive oil the primary fat.
  Interventions: Drug: Metformin; Drug: GLP-1A; Dietary Supplement: MED

INTERVENTIONS:
Drug: Metformin — 16 weeks of using metformin: Dosing will initiate at 500mg TID and increased to 1000mg BID after one week.
  Other Names: MET
Drug: GLP-1A — 16 weeks using GLP1a: Dosing will be titrated per clinical guidelines and as per FDA approved clinical protocols.
  Other Names: Glucagon-like peptide-1 analog
Dietary Supplement: MED — 16 weeks of following a Mediterranean diet: a mostly plant-based diet that includes vegetables, whole grains, whole fruits, legumes, nuts and seeds, with fish being the primary animal protein, and olive oil the primary fat.
  Other Names: Mediterranean Diet; energy-restricted Mediterranean diet

SUMMARY:
The study team will invite participants with prediabetes or mild diabetes (HbA1c 5.7-7.0) to join a 5-year research study that will define subphenotypes of type 2 diabetes based on underlying physiology (eg insulin resistance, beta-cell dysfunction, incretin defect, liver insulin resistance) and then test the hypothesis that response to three first-line treatments will vary according to metabolic subphenotype. Variables of interest include glucose, cardiovascular risk markers, and weight. Treatments include Mediterranean diet, metformin, and a GLP-1 agonist. Participants will go through an initial screening, followed by three treatment periods, each lasting 4 months with 3 month washout in-between treatment periods. This study will help us understand how personalized treatments can help control blood glucose, reduce cardiovascular risk, and manage weight. While there may be minor side effects-like slight discomfort from blood tests, gastrointestinal symptoms from some of the medications, and small radiation exposure from DXA body scans-the treatments offered in this study have all been well studied and are known to lower risk for diabetes and cardiovascular disease

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥23 (≥22 in Asians) kg/m2 but < 45 kg/m2
* HbA1c 5.7-8.0% while not on antihyperglycemic medications

Exclusion Criteria:

* Recent (<6mos) CVD event
* active malignancy, kidney/liver disease pregnancy/lactation, chronic inflammatory disease, eating disorder, bariatric surgery
* history of acute pancreatitis
* family or personal history of medullary thyroid cancer
* current use of antihyperglycemic, diabetogenic, or weight loss medications (washout allowed if approved by primary physician)
* heavy alcohol use
* hct <30, creatinine > 1.4, ALT> 3x ULN
* physical activity >2 hours/day
* inability to come to Stanford CTRU for metabolic testing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | At month 0, month 4, month 8, month 11, month 15, month 18
  The study team will compare the change in HbA1c levels from beginning to end of intervention to compare the efficacy of each treatment.

SECONDARY OUTCOMES:
Change in Time in Range (TIR) | At month 0, month 4, month 8, month 11, month 15, month 18
  Change in Time in Rage (TIR) as measured by continuous glucose monitor (CGM). TIR is defined as a range of 70-140 mg/dL. The study team will calculate the changes from beginning to end or each intervention and compare efficacy of each treatment in TIR.
Change in body weight | At month 0, month 4, month 8, month 11, month 15, month 18
  Compare efficacy of each treatment in change in body weight (kg).
Change in Blood Pressure | At month 0, month 4, month 8, month 11, month 15, month 18
  Compare efficacy of each treatment in change in blood pressure.
Change in LDL Cholesterol | At month 0, month 4, month 8, month 11, month 15, month 18
  Change in LDL cholesterol at the beginning and end of each intervention to compare the efficacy of each treatment.
Change in Triglycerides | At month 0, month 4, month 8, month 11, month 15, month 18
  Change in triglycerides at the beginning and end of each intervention period to compare the efficacy of each treatment.
Change in high-sensitivity C-reactive protein (hsCRP) | At month 0, month 4, month 8, month 11, month 15, month 18
  hsCRP will be measured at the beginning and end of each intervention period to compare the efficacy of each treatment.
Change in alanine transaminase (ALT) | At month 0, month 4, month 8, month 11, month 15, month 18
  ALT will be measured at the beginning and end of each intervention period to compare the efficacy of each treatment.
Change in adiponectin | At month 0, month 4, month 8, month 11, month 15, month 18
  Adiponectin will be measured at the beginning and end of each intervention period to compare the efficacy of each treatment.
HOMA-B | At month 0, month 4, month 8, month 11, month 15, month 18
  Change from baseline in HOMA-B at the beginning and end of each intervention period to compare the efficacy of each treatment.
HOMA-IR | At month 0, month 4, month 8, month 11, month 15, month 18
  Change from baseline in HOMA-IR at the beginning and end of each intervention period to compare the efficacy of each treatment.
Change in body fat mass | At month 0, month 4, month 8, month 11, month 15, month 18
  Body fat mass will be measured by dual-energy x-ray absorptiometry (DXA) scan at the beginning and end of each intervention period to compare the efficacy of each treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Tracey McLaughlin, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No